CLINICAL TRIAL: NCT05856786
Title: To Study the Effects of Refractive Surgery on Optical Coherence Tomography (OCT) Measurements in the Eye: A Pilot Study
Brief Title: To Study the Effects of Refractive Surgery on OCT Measurements in the Eye
Status: Recruiting | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0262-22-EP
Record Dates: First submitted 2023-04-24; First posted 2023-05-12 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Optical Coherence Tomography; Refractive Errors; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ocular parameters: Patients aged 19 years or more who are scheduled to undergo refractive surgery will be included in the study. OCT will be performed at baseline (before surgery), 1 day after surgery and 1 week after surgery. Each patient will be tested 3 times.
  Interventions: Diagnostic Test: Optical coherence tomography

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography — Posterior segment OCT (a non-contact procedure performed over one minute) is additionally performed for patients participating in this study. Proportion of change in measurements in microns will be analyzed.

SUMMARY:
Corrective eye surgeries, such as Lasik, are widely used to correct focusing problems such as myopia, or nearsightedness. Often these patients develop other conditions like myopic maculopathy or glaucoma which require monitoring with optical coherence tomography (OCT). Since OCT is a light-based test and changes the refractive status of the eye (in the cornea or the lens), it can potentially affect the results of the OCT measurements but has not been sufficiently studied. This pilot study aims at studying the potential change in OCT parameters in the eye after undergoing such surgery.

DETAILED DESCRIPTION:
Refractive surgeries are widely used in patients with ametropia. Refractive surgery is most commonly performed in patients with myopia. These patients often have a predilection for developing other conditions in the posterior segment of the eye, like myopic maculopathy or glaucoma which require monitoring with optical coherence tomography (OCT). Since OCT is a light-based test and changes in the refractive status of the eye (in the cornea or the lens) can potentially affect the results of the OCT measurements. Literature review reveals that the effect of significant changes in refractive power of the eye on the parameters of optical coherence tomography (OCT) has not been sufficiently studied. Some authors simulated the effect of refractive surgery using a contact lens but had diverging results. This prospective pilot study aims at studying the potential change in OCT parameters in the eye after undergoing refractive surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing refractive surgery
2. For patients undergoing bilateral eye surgery, the one with higher degree of ametropia will be included.

Exclusion Criteria:

1. Astigmatism more than 3 Diopters
2. Visual acuity worse than 20/25
3. Patients with unstable visual fixation
4. Severe Dry Eye

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All subjects in the study will be adults aged 19 years or more, that fits the typical age profile of patients in the refractive surgery clinic. Refractive surgery is an elective surgery and the patients are encouraged to ask questions about the study. This is an observational study and all aspects of care, including procedures, visits, and exams, carried out as part of the study represent standard of care. Patients visiting the refractive surgery clinic will be given an option to participate in the study if they meet the selection criteria. The clinical care of the patient will not be affected by the patient's participation or non-participation in the study.
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Macular thickness | 1 day after refractive procedure
  Proportion of Change in thickness of retina and its layers measured in microns
Macular thickness | 1 week after refractive procedure
  Proportion of Change in thickness of retina and its layers measured in microns

SECONDARY OUTCOMES:
Choroidal thickness | 1 day after refractive procedure
  Proportion of Change in thickness of choroid and its layers measured in microns
Choroidal thickness | 1 week after refractive procedure
  Proportion of Change in thickness of choroid and its layers measured in microns
visual acuity | 1 day after refractive procedure
  Proportion of Change in clarity of vision, measured in logarithm of Minimal Angle of Resolution (logMAR) units
visual acuity | 1 week after refractive procedure
  Proportion of Change in clarity of vision, measured in logarithm of Minimal Angle of Resolution (logMAR) units
central corneal thickness | 1 day after refractive procedure
  Proportion of Change in thickness of cornea measured in microns
central corneal thickness | 1 week after refractive procedure
  Proportion of Change in thickness of cornea measured in microns
anterior chamber depth | 1 day after refractive procedure
  Proportion of Change in depth of anterior chamber of the eye measured in microns
anterior chamber depth | 1 week after refractive procedure
  Proportion of Change in depth of anterior chamber of the eye measured in microns
keratometry | 1 day after refractive procedure
  Proportion of Change in corneal curvature measured in diopters
keratometry | 1 week after refractive procedure
  Proportion of Change in corneal curvature measured in diopters

CONTACTS AND LOCATIONS:
Overall Officials: Pukhraj P Rishi, MBBS, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Y, Liao H, Sun Y, Shen X. Short-term changes in the anterior segment and retina after small incision lenticule extraction. BMC Ophthalmol. 2020 Oct 7;20(1):397. doi: 10.1186/s12886-020-01668-7. PMID 33028265
- [Background] Shpak AA, Kostenev SV, Mushkova IA, Korobkova MV. [Effect of corneal refractive surgery on optical coherence tomography measurements]. Vestn Oftalmol. 2018;134(5):48-53. doi: 10.17116/oftalma201813405148. Russian. PMID 30499539
- [Background] Ozsaygili C, Altunel O, Duru N. Evaluation of the change in retinal thickness after femtosecond laser-assisted laser in situ keratomileusis and photorefractive keratectomy. Curr Eye Res. 2022 Jan;47(1):18-24. doi: 10.1080/02713683.2021.1951297. Epub 2021 Jul 7. PMID 34231433
- [Background] Yalcinkaya G, Yildiz BK, Cakir I, Yildirim Y, Demirok A. Evaluation of peripapillary - macular microvascularity and choroidal vascularity index after refractive surgery. Photodiagnosis Photodyn Ther. 2022 Mar;37:102714. doi: 10.1016/j.pdpdt.2022.102714. Epub 2022 Jan 5. PMID 34995787